CLINICAL TRIAL: NCT03749382
Title: A Randomized Controlled Trial of Smoking Interventions in Women
Brief Title: Testing Smoking Interventions in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Lucy Walker, Prinical Investigator, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0245
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Smoking Cessation
Keywords: Smoking; Tobacco; Cessation; Intervention
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Smoking Devices

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant
Masking Description: Participants will receive a brief description of both the appearance-based intervention and general stop smoking intervention. Participants will not know prior to taking part which condition they will be randomised into, on completion of the intervention it will become apparent whether they received the appearance-based intervention or general intervention. For participants randomised to the appearance intervention the instruction type will remain concealed. The investigator will not be blind throughout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Neutral instructions (Experimental): Appearance based intervention group delivered with neutral instructions from the investigator alongside general stop smoking intervention leaflet.
  Interventions: Other: AprilAge- facial morphing appearance based intervention for smoking
- Intervention Additional instructions (Experimental): Appearance based intervention group delivered with neutral instructions with additional reassuring messages from the investigator alongside general stop smoking intervention leaflet.
  Interventions: Other: AprilAge- facial morphing appearance based intervention for smoking
- Control (No Intervention): Neutral task plus the general stop smoking intervention in the form of a leaflet, administered by the investigator.

INTERVENTIONS:
Other: AprilAge- facial morphing appearance based intervention for smoking — Appearance-based intervention: The intervention is a software that ages an individual's face with and without the effects of smoking. Participants have their photo taken on a laptop webcam, they are then asked to report their age and ethnicity in order to calibrate the software, the participants picture is then matched to a stock image. The participants will see two images on the screen, on the left is there face aged without the effects of smoking and one the right aged with the effects of smoking. Participants will be led through a series of morphing sequences (1-5). In-between each of the morphing sequences (Morph1 to Morph5) the participant will be asked to comment on the differences they can see between the two images.
  General stop smoking intervention: The General stop smoking intervention comes in the form of a NHS stop smoking information leaflet. The participants will be given the leaflet on a laptop screen and asked to read through the whole document.
  Other Names: Appearance-based intervention; Appearance orientated intervention; Internet-based Photo aging intervention
  Arms: Intervention Additional instructions; Intervention Neutral instructions

SUMMARY:
The study is a randomised controlled trial (RCT) designed to test two tailored conditions of an appearance-based intervention for smoking in female smokers, compared to a control group administered a general stop smoking intervention.

The intervention delivery is being tested to assess whether the level of physiological arousal evoked by the intervention and the instruction type has an influence on the outcome measures. To do this one condition will receive the intervention with a neutral instruction and the other the intervention with additional instructions, measures of physiological stress reactivity will be used to measure level of stress evoked by the intervention and delivery.

DETAILED DESCRIPTION:
Background

Despite health-related smoking cessation campaigns, still one in five of adults in the UK smokes and it is estimated that half of all regular smokers will eventually die from smoking-related diseases. Innovative smoking cessation campaigns are needed to reach the remaining smoker population and prevent smoking-related diseases.

Smoking interventions have previously focused on smoking impact on health. However, besides health-related diseases, smoking causes aging effects to the skin and recent research suggests that smoking interventions based on threats to appearance may be more effective. Further research using an age-appearance facial morphing intervention for smoking, which shows women realistic images of the effects of smoking on their own face, research found that female smokers aged 18-34 reported increased motivation to quit after the intervention. Quantitative results from a randomised control trial support the interventions effectiveness .

The previous research on appearance-based interventions for smoking show promising results however these studies had report small sample sizes and differences in the age range of participants. Additionally, previous research has focused on the primary outcome measures of smoking including smoking cognitions, behaviours and CO readings and have not investigated further moderating variables such as, anxiety, depression, appearance orientation and stage of change.

In previous research participants have consistently reported a 'shock' reaction, and findings from a pilot and feasibility study (unpublished) suggest that this 'shock' reaction as measured by physiological reactivity to the intervention could mediate smoking outcomes. Therefore, the present research proposes to assess facial morphing intervention effectiveness in relation to individual's physiological shock reactions to viewing the morphed images and moderator variables in a large sample of women across a broad age range.

Objectives:

Primary Objectives- To assess effectiveness of an appearance-based intervention on smoking outcomes in a female population (18-55 years old) immediately after the intervention session and at 1, 3 and 6 months post intervention session. In addition to compare the results to that of a standard stop smoking intervention.

An additional primary objective will be to compare the primary outcome measures for both appearance-based intervention instruction conditions (neutral vs additional) immediately after the intervention and at 1, 3 and 6 months after to assess which instruction type is more effective in reducing smoking behaviour.

Other objectives-

1. Investigate the mediating effects of physiological arousal [measured during the intervention by electro dermal activity and beats per a minute (BPM, derived from pulse rate)] on the intervention efficacy as measured by the primary and secondary outcome measures.
2. Investigate the impact of moderating variables on the primary outcome measures.

Measures

Outcome measures -

1. The primary outcomes will be smoking intentions measured pre, immediately after and at 1, 3 and 6 months post intervention.
2. Secondary outcome measures will be smoking cognitions (attitudes, subjective norms and perceived behavioural control), nicotine dependence and self-reported smoking behaviour measured pre, immediately after and at 1, 3 and 6 month post the intervention.

Participants:

Current female smokers aged 18-55 will be recruited and randomised into one of three conditions. (1) Appearance-based intervention neutral, (2) Appearance-based intervention additional instructions, (3) Control general stop smoking intervention. Participants are eligible to take part if they are a female between the ages of 18-55 and that they smoke at least one cigarette a week. Participants are informed to withhold from taking part if they have any mental health issues that may be affected by appearance-based imagery.

Randomisation will be achieved through using SPSS (V25) to create two sets of randomisation one for participants over the age of 35 and another for women under the age 35 to allow an equal distribution of ages into each condition.

Protocol:

At the start of the intervention session participants will be asked to provide informed consent, immediately after electrodes and a light sensor will be placed on the participants non-dominant hand. Participants are then asked to fill in a self-report questionnaire including demographic questions and stress confounders, smoking behaviour, cognitions and quit attempts, levels of anxiety and depression, how much they consider their future consequences and how they view their appearance.

Participants in the two appearance-based interventions groups will then have a photo taken of their face and aged with the effects of smoking in a range of morphing sequences and then given a general stop smoking booklet alternatively participants allocated to the control condition will be asked to only read a general stop smoking intervention booklet. All three conditions will then be asked to provide carbon monoxide breath reading using a hand held battery operated device. The participants smoking cognitions and behaviours will then be measured again immediately and longer term at 1, 3 and 6 months post intervention.

Sample size calculation:

In a previous randomized controlled trial (RCT) on an appearance-based intervention for female smokers , 35 women were allocated to one of two conditions (control group or intervention) with a reported effect size of d=.63 for nicotine dependence at 4 weeks post-intervention. Based on previous research and to account for a 30% dropout at six-month follow up 50 participants per group is required in the current study. Additionally, an a priori power analysis has been conducted using GPower which supports the specified number of participants per group. Specifically, to obtain a medium effect of .25 and a power of .80 at alpha .05, a total sample of 158 is required (52 per group).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-55
* Smoke at least 1 cigarette a week

Exclusion Criteria:

* Non-smokers
* Self-reported appearance related mental health issue

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Smoking Intentions | Measure obtained pre-intervention, immediately after the intervention and again at 1, 3 and 6 months post-intervention.
  Smoking Intentions, which are intentions the participant has to quit smoking are measured via self-report as part of the Smoking Questionnaire (Grogan et al., 2011) based on the theory of planned behaviour construct (Ajzen, 1991). Three items are each asked on a 13-point scale producing a combined score between 0-39. The score from each individual item is then averaged together to create a total score for smoking intentions. The higher the averaged score the more intention the participant has to quit smoking.The scale has previously been used in similar appearance-based interventions for smoking research (Grogan et al., 2011).

SECONDARY OUTCOMES:
Change in Smoking Attitudes | Measures obtained pre-intervention, immediately after the intervention and again at 1, 3 and 6 months post-intervention.
  Smoking Attitudes, is the attitude a participant has to smoking cessation, measured via self-report as part of the Smoking Questionnaire (Grogan et al., 2011) based on the theory of planned behaviour construct (Ajzen, 1991). Four items are each asked on a 13-point scale producing a score between 0-52. Scores from individual items are then averaged together to create a total score for Smoking Attitudes. The higher the averaged score the more positive the participants attitude is to smoking cessation. The scale has previously been used in similar appearance-based interventions for smoking research (Grogan et al., 2011).
Change in Smoking Subjective Norms | Measure obtained pre-intervention, immediately after the intervention and again at 1, 3 and 6 months post-intervention.
  Smoking Subjective Norms, is the perceived social pressure the participant feels to stop smoking, measured via self-report as part of the Smoking Questionnaire (Grogan et al., 2011) based on the theory of planned behaviour construct (Ajzen, 1991). Three items are each asked on a 13-point scale producing a combined score between 0-39. Scores from each individual item is then averaged together to create a total score for Smoking Subjective Norms. The higher the averaged score the more the participants feels it socially acceptable to quit smoking .The scale has previously been used in similar appearance-based interventions for smoking research (Grogan et al., 2011).
Change in Smoking Perceived Behavioural Control | Measure obtained pre-intervention, immediately after the intervention and again at 1, 3 and 6 months post-intervention.
  Smoking Subjective Perceived Behavioural Control, is the Perceived Control the participant has over their own smoking behaviour, measured via self-report as part of the Smoking Questionnaire (Grogan et al., 2011) based on the theory of planned behaviour construct (Ajzen, 1991). Four items are each asked on a 13-point scale producing a combined score between 0-52. Scores from each individual item is then averaged together to create a total score for Smoking Perceived Behavioural Control. The higher the averaged score the more control a participants feels they have over their own smoking behaviour. The scale has previously been used in similar appearance-based interventions for smoking research (Grogan et al., 2011).
Change in Nicotine dependence | Measure obtained pre-intervention and again at 1, 3 and 6 months post-intervention.
  Nicotine dependence as measured by the Fagerstrom test for nicotine dependence (Heatherton et al.,1991) a validated instrument that determines the extent to which participants are physically addicted to nicotine. The measure includes six items that are summed to create a score between 0-10. Higher scores equate to a higher dependence to nicotine.
Change in Self-reported smoking behaviour | Measure obtained pre-intervention and again at 1, 3 and 6 months post-intervention.
  Participants report the amount of cigarettes smoked each day for the week prior to each measurement time point, the cigarettes consumed on each day are summed to create a total cigarette consumption score for the week. The measure is administered to the participant as part of the Smoking Questionnaire (Grogan et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Brooks Building, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Borrelli B, Mermelstein R. The role of weight concern and self-efficacy in smoking cessation and weight gain among smokers in a clinic-based cessation program. Addict Behav. 1998 Sep-Oct;23(5):609-22. doi: 10.1016/s0306-4603(98)00014-8. PMID 9768298
- [Background] Cash, T. F. (2016) 'Multidimensional Body-Self Relations Questionnaire (MBSRQ).' In Wade, T. (ed.) Encyclopedia of Feeding and Eating Disorders. Singapore: Springer Singapore, pp. 1-4.
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Flett K, Clark-Carter D, Grogan S, Davey R. How effective are physical appearance interventions in changing smoking perceptions, attitudes and behaviours? A systematic review. Tob Control. 2013 Mar;22(2):74-9. doi: 10.1136/tobaccocontrol-2011-050236. Epub 2012 May 9. PMID 22573734
- [Background] Flett K, Grogan S, Clark-Carter D, Gough B, Conner M. Male smokers' experiences of an appearance-focused facial-ageing intervention. J Health Psychol. 2017 Mar;22(4):422-433. doi: 10.1177/1359105315603477. Epub 2016 Jul 10. PMID 26338489
- [Background] Grogan S, Flett K, Clark-Carter D, Gough B, Davey R, Richardson D, Rajaratnam G. Women smokers' experiences of an age-appearance anti-smoking intervention: a qualitative study. Br J Health Psychol. 2011 Nov;16(4):675-89. doi: 10.1348/2044-8287.002006. Epub 2010 Dec 6. PMID 21199543
- [Background] Grogan S, Flett K, Clark-Carter D, Conner M, Davey R, Richardson D, Rajaratnam G. A randomized controlled trial of an appearance-related smoking intervention. Health Psychol. 2011 Nov;30(6):805-9. doi: 10.1037/a0024745. Epub 2011 Jul 18. PMID 21767016
- [Background] Gupta SK. Intention-to-treat concept: A review. Perspect Clin Res. 2011 Jul;2(3):109-12. doi: 10.4103/2229-3485.83221. PMID 21897887
- [Background] Koh JS, Kang H, Choi SW, Kim HO. Cigarette smoking associated with premature facial wrinkling: image analysis of facial skin replicas. Int J Dermatol. 2002 Jan;41(1):21-7. doi: 10.1046/j.1365-4362.2002.01352.x. PMID 11895509
- [Background] Strathman, A., Gleicher, F., Boninger, D. S. and Edwards, C. S. (1994) 'The consideration of future consequences: Weighing immediate and distant outcomes of behavior.' Journal of Personality and Social Psychology, 66(4) pp. 742-752.
- [Derived] Walker L, Grogan S, Denovan A, Scholtens K, McMillan B, Conner M, Epton T, Armitage CJ, Cordero MI. An Age-Progression Intervention for Smoking Cessation: A Pilot Study Investigating the Influence of Two Sets of Instructions on Intervention Efficacy. Int J Behav Med. 2024 May 9. doi: 10.1007/s12529-024-10285-3. Online ahead of print. PMID 38724879